CLINICAL TRIAL: NCT01166425
Title: A Randomized, Double-blind, Placebo Controlled Study of the Efficacy of Lithium for the Treatment of Pediatric Mania Followed by an Open Label Long-term Safety Period, Double-blind, Placebo-controlled Discontinuation Phase, and Open Label Restabilization Period.
Brief Title: Safety and Efficacy Study of Lithium for the Treatment of Pediatric Mania.
Acronym: Lithium2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-2005-07-2
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-05

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium Carbonate; Lithium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium Carbonate (Active Comparator): Participants weighing ≥ 30 kg who are randomized to receive active lithium will begin treatment at 300 mg TID (three times a day) at visit 1 (total dose 900 mg). Participants weighing < 30 kg who are randomized to receive active lithium will begin treatment at 300 mg BID (two times a day) the day after visit 1 (total dose 600 mg). Based on the participant's response and tolerability, the dose will be increased by 300mg three days after the baseline visit and at scheduled in-office visits to the maximum tolerated dose.
  Interventions: Drug: Lithium Carbonate
- placebo (Placebo Comparator): Participants who are randomized to receive placebo during the Efficacy Phase will receive matching placebo capsules. Dosing will be titrated as described for active lithium.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium Carbonate — Participants weighing ≥ 30 kg who are randomized to receive active lithium will begin treatment at 300 mg TID at visit 1 (total dose 900 mg). Participants weighing < 30 kg who are randomized to receive active lithium will begin treatment at 300 mg BID the day after visit 1 (total dose 600 mg). Based on the participant's response and tolerability, the dose will be increased by 300mg three days after the baseline visit and at scheduled in-office visits to the maximum tolerated dose. One mid-week dose increase will be scheduled in addition to the weekly increases at the scheduled in-clinic visits. On day 3 (+/- 2 days), a dose increase of 300 mg may occur based on the results of a telephone call placed by the study investigator to the participant's parent/guardian. During the telephone call, the prescribing clinician will assess medication adherence, adverse events, and overall improvement since baseline.
  Other Names: Lithium capsules
  Arms: Lithium Carbonate
Drug: Placebo — Participants who are randomized to receive placebo during the Efficacy Phase will receive matching placebo capsules. Dosing will be titrated as described for active lithium.
  Other Names: Placebo capsules
  Arms: placebo

SUMMARY:
Study Design This is the second study of a multiphase, multicenter trial that will comprehensively examine lithium in the treatment of pediatric participants with bipolar I disorder. In order to examine the treatment of bipolar disorder with lithium, this study will include four phases of treatment. The first phase, the Efficacy Phase, will include participants being randomized to either lithium or placebo for 8 weeks to determine the efficacy of lithium in the treatment of children and adolescents with bipolar I disorder. Once participants complete the Efficacy Phase, participants may be eligible to continue in the Long- Term Effectiveness Phase for a maximum of 24 weeks of lithium treatment. Subsequently, participants meeting response criteria during the Long-Term Effectiveness Phase will be eligible to continue in the Discontinuation Phase. During the Discontinuation Phase, participants will be randomized to either placebo or lithium treatment for up to 28 weeks. Finally, those participants who experience a mood relapse during the Discontinuation Phase will be enrolled in an Open Label Restabilization Phase and treated with lithium for up to 8 weeks.

DETAILED DESCRIPTION:
The following are the objectives of this study:

1. To determine if lithium is more efficacious in reducing symptoms of mania than placebo.
2. To describe the short-term safety of lithium in the pediatric population relative to placebo treatment.
3. To examine the effectiveness and efficacy of lithium as a maintenance treatment for children and adolescents with bipolar I disorder.
4. To examine the long-term and short-term safety and tolerability of lithium in pediatric bipolar I disorder.
5. To examine the effects of lithium treatment over time on specific aspects of cognitive functioning that have been reported to be adversely affected by lithium in the adult population.
6. More specifically, to determine the integrity of fine-motor, attention, verbal memory, and selected executive function domains prior to treatment at baseline, at the end of week 8/early termination of the Efficacy Phase, and at the end of week 24/early termination from the Long- Term Effectiveness Phase (after 24/32 weeks of lithium treatment).
7. To examine the relationship between systemic exposure to lithium and effectiveness and toxicity.
8. To examine the long-term safety and tolerability of combination therapy, lithium plus other psychotropic agents, in pediatric bipolar I disorder.
9. To critically assess the efficacy of lithium for prophylaxis against recurrence of mood symptoms in children and adolescents.
10. In those participants who discontinue treatment with lithium and experience a mood relapse, to determine the duration of lithium treatment necessary before re-stabilization is achieved.
11. To evaluate the influence of intrinsic factors [e.g. age, gender, race, renal function, height, (measured by stadiometer) and weight] on lithium exposure.

The Study population for this study: Children and adolescents 7- 17 years of age who meet DSM-IV diagnostic criteria for Bipolar I (mania, mixed mania) without psychotic symptoms as determined by a child and adolescent psychiatrist will be eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 7 years to 17 years, 11 months old at time of first dose
2. Participants must meet DSM-IV diagnostic criteria, as assessed by a semi-structured assessment (KSADS-PL) and a separate clinical interview with a child/adolescent psychiatrist for manic or mixed episodes in bipolar I disorder
3. Score of > 20 on the YMRS at screening and baseline
4. The participant and legal guardian must understand the nature of the study and be able to comply with protocol requirements. The legal guardian must give written informed consent and the youth, written assent
5. Participants with comorbid conditions [attention deficit hyperactivity disorder (ADHD), conduct disorder], except those listed in Exclusion Criterion 2, may participate
6. If female: is premenarchal, or is incapable of pregnancy because of a hysterectomy, tubal ligation, or spousal/partner sterility. If sexually active and capable of pregnancy, has been using an acceptable method of contraception (hormonal contraceptives, intrauterine device, spermicide and barrier) for at least one month prior to study entry and agrees to continue to use one of these for the duration of the study. If sexually abstinent and capable of pregnancy, agrees to continued abstinence or to use of an acceptable method of birth control should sexual activity commence
7. Has a negative quantitative serum ß-human chorionic gonadotrophin hormone pregnancy test at screening and a negative qualitative urine pregnancy test at baseline, if female
8. Participants with a history of substance abuse may participate if they agree to continue to abstain from drugs during the trial and have a negative drug screen at screening or prior to baseline. Those with an initial positive drug screen during screening may have another screen done 1-3 weeks later while in screening, and a negative result will allow the participant to participate
9. The participant is willing and clinically able to wash out of exclusion medications during the screening period. Prior to the administration of lithium, participants will have not used any of the following medications: antipsychotics, monoamine oxidase inhibitors, antidepressants within the preceding 2 weeks; stimulants within the preceding week; or fluoxetine or depot antipsychotics in the past month (no stable participants will be asked to discontinue medications)
10. ECG and bloodwork including CBC, electrolytes, etc. (as per Safety assessment procedures listed in Table 6) showing no clinically significant abnormalities

Exclusion Criteria:

1. Participant who is clinically stable on current medication regimen for bipolar disorder
2. A current or lifetime diagnosis of Schizophrenia or Schizoaffective Disorder, a Pervasive Developmental Disorder (ASQ score > 15), Anorexia Nervosa, Bulimia Nervosa, or Obsessive-Compulsive Disorder
3. Current DSM-IV diagnosis of Substance Dependence
4. Positive drug screen at screening and on retest 1-3 weeks later
5. Participants with symptoms of mania that may be attributable to a general medical condition, or secondary to use of medications (e.g., corticosteroids)
6. Evidence of any serious, unstable neurological illness for which treatment under the auspices of this study would be contraindicated
7. Any serious, unstable medical illness or clinically significant abnormal laboratory assessments that would adversely impact the scientific interpretability or unduly increase the risks of the protocol
8. Current general medical condition including neurological disease, diabetes mellitus, thyroid dysfunction, or renal dysfunction that might be affected adversely by lithium, could influence the efficacy or safety of lithium, or would complicate interpretation of study results
9. Evidence of current serious homicidal/suicidal ideation such that in the treating physician's opinion it would not be appropriately safe for the participant to participate in this study
10. Evidence of current active hallucinations and delusions such that in the treating physician's opinion it would not be appropriately safe for the participant to participate in this study
11. Concomitant prescription of over-the-counter medication or nutritional supplements (e.g., ibuprofen, naproxen, St John's wort) that would interact with lithium or affect the participant's physical or mental status
12. Concomitant psychotherapy treatments provided outside the study initiated within 4 weeks prior to screening
13. Previous adequate trial with Li+ (at least 4 weeks with Li+ serum levels between 0.8-1.2 mEq/L)
14. History of allergy to lithium or lithium intolerance
15. Psychiatric hospitalization within 1 month of screening for psychosis or serious homicidal/serious suicidal ideation
16. Clinician's judgment that participant is not likely to be able to complete the study as an outpatient due to psychiatric reasons
17. Females who are currently pregnant or lactating
18. Sexually active females who, in the investigators' opinion, are not using an adequate form of birth control.
19. Participants who are unable to swallow the study medication
20. Participants for whom a baseline YMRS score of < 20 is anticipated
21. Participants with an IQ less than 70 (determined using the Wechsler Abbreviated Scales of Intelligence {WASI} Vocabulary and Matrix Reasoning Subscales)

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2010-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
YMRS score | >17 months
  Significant changes in YMRS scores from baseline to the end of each study phase.
  YMRS scores are questionnaires to assess pediatric mania.

SECONDARY OUTCOMES:
Clinical Global Impressions Scale- Severity and Improvement | >17 months
Children Depression Rating Scale-Revised | >17 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Findling, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (11):
- United States (11):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - University of Illinois at Chicago, South Chicago Heights, Illinois
  - University of Kansas School of Medicine, Psychiatry and Behavioral Sciences, 1010 N Kansas St, Wichita, Kansas
  - University of Massachusetts Medical School, Biotech One Suite 100, 365 Plantation, Worcester, Massachusetts
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Department of Psychiatry, CB 7160, Chapel Hill, North Carolina
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Seattle Childrens Hospital Research Institute, Seattle, Washington

REFERENCES:
- [Derived] Findling RL, McNamara NK, Pavuluri M, Frazier JA, Rynn M, Scheffer R, Kafantaris V, Robb A, DelBello M, Kowatch RA, Rowles BM, Lingler J, Zhao J, Clemons T, Martz K, Anand R, Taylor-Zapata P. Lithium for the Maintenance Treatment of Bipolar I Disorder: A Double-Blind, Placebo-Controlled Discontinuation Study. J Am Acad Child Adolesc Psychiatry. 2019 Feb;58(2):287-296.e4. doi: 10.1016/j.jaac.2018.07.901. Epub 2018 Nov 26. PMID 30738555
- [Derived] Findling RL, Robb A, McNamara NK, Pavuluri MN, Kafantaris V, Scheffer R, Frazier JA, Rynn M, DelBello M, Kowatch RA, Rowles BM, Lingler J, Martz K, Anand R, Clemons TE, Taylor-Zapata P. Lithium in the Acute Treatment of Bipolar I Disorder: A Double-Blind, Placebo-Controlled Study. Pediatrics. 2015 Nov;136(5):885-94. doi: 10.1542/peds.2015-0743. Epub 2015 Oct 12. PMID 26459650